CLINICAL TRIAL: NCT05732376
Title: Investigation of the Effectiveness of Simulation-Based Functional Nasopharyngoscopic Velopharyngeal Assessment Trainings Given to Speech and Language Therapy Students
Brief Title: Effectiveness of Two Simulation-Based Functional Nasopharyngoscopic Velopharyngeal Assessment Trainings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Namık Yücel Birol, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEDIPOL-SLT-BIROL-001
Record Dates: First submitted 2023-01-28; First posted 2023-02-17 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Simulation Training
Keywords: simulation; nasopharyngoscopy training; speech and language therapy
MeSH Terms: conditions — Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D Printed Endoscopy Training Model Group (Experimental)
  Interventions: Behavioral: Nasopharyngoscopic Velopharyngeal Training with 3D Printed Endoscopy Training Model
- Ready-Made Endoscopy Training Model Group (Active Comparator)
  Interventions: Behavioral: Nasopharyngoscopic Velopharyngeal Training with Ready-Made Endoscopy Training Model

INTERVENTIONS:
Behavioral: Nasopharyngoscopic Velopharyngeal Training with 3D Printed Endoscopy Training Model — Theoretical training: The theoretical training covers the anatomy and physiology of the velopharyngeal region and nasal cavity, nasopharyngoscope, preparation of the patient for nasopharyngoscopy, use of the endoscope during nasopharyngoscopy and the procedure for nasopharyngoscopic velopharyngeal function assessment.
  Practical training: At the beginning of the hands-on training, the device will be introduced to the participants. Basic information will be given about endoscopy device. Then, the principal investigator will give information about the use of the endoscope (patient instructions, holding the endoscope, placement of the endoscope in the nose, manipulation of the endoscope, anatomical structures in the nasal cavity and velopharyngeal region, velopharyngeal function assessment) on the 3D printed endoscopy training model. Participants will receive hands-on training on the 3D printed endoscopy training model, under the guidance of the principal investigator.
  Arms: 3D Printed Endoscopy Training Model Group
Behavioral: Nasopharyngoscopic Velopharyngeal Training with Ready-Made Endoscopy Training Model — Theoretical training: The theoretical training covers the anatomy and physiology of the velopharyngeal region and nasal cavity, nasopharyngoscope, preparation of the patient for nasopharyngoscopy, use of the endoscope during nasopharyngoscopy and the procedure for nasopharyngoscopic velopharyngeal function assessment.
  Practical training: At the beginning of the hands-on training, the device will be introduced to the participants. Basic information will be given about endoscopy device. Then, the principal investigator will give information about the use of the endoscope (patient instructions, holding the endoscope, placement of the endoscope in the nose, manipulation of the endoscope, anatomical structures in the nasal cavity and velopharyngeal region, velopharyngeal function assessment) on the ready-made endoscopy training model. Participants will receive hands-on training on the ready-made endoscopy training model, under the guidance of the principal investigator.
  Arms: Ready-Made Endoscopy Training Model Group

SUMMARY:
The aim of this clinical trial was to compare the effectiveness of functional nasopharyngoscopic velopharyngeal assessment training given to undergraduate speech and language therapy students on a 3D printed endoscopy training model and a ready-made endoscopy training model.

ELIGIBILITY:
Inclusion Criteria:

* To be a 4th year undergraduate student of speech and language therapy
* To have taken the course of cleft lip and palate or an equivalent course

Exclusion Criteria:

* Receiving previous hand-on flexible endoscopy training
* Having any health problem in the upper extremities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Nasopharyngoscopic Velopharyngeal Evaluation Clinician Experience | 2 Months
  A 9-question perceptual survey was created to evaluate the participants' self-confidence and self-competence in performing nasopharyngoscopic velopharyngeal evaluation. The survey was adapted from a 5-point Likert-type survey previously used in simulation-based transnasal endoscopy training on swallowing assessment (Benadom & Potter, 2011).

SECONDARY OUTCOMES:
Procedure time | 2 Months
  This is the time from the moment the endoscope enters the nostril until it reaches the point of visualization of the velopharyngeal sphincter. This time does not include the time the endoscope is removed from the nose and reinserted.
Volunteer Experience for Nasopharyngoscopic Velopharyngeal Evaluation | 2 Months
  A 6-question survey was created to allow volunteers to perceptually assess the competence and confidence of the clinician after the endoscope was administered to the volunteers. The survey was adapted from a 5-point Likert-type survey previously used in simulation-based transnasal endoscopy training in swallowing assessment (Benadom & Potter, 2011).
Training Satisfaction Survey | 2 Months
  A training satisfaction survey consisting of a total of 7 questions (four Likert-type and three open-ended question) was created to learn the evaluations of the participants regarding the importance, effectiveness, appropriateness and satisfaction level of the simulation trainings. The survey was adapted from the form created by Uz-Hasırcı (2020).

CONTACTS AND LOCATIONS:
Overall Officials: Namık Y. Birol, Doctoral Student, Principal Investigator — Istanbul Medipol University, Institute of Health Sciences, Department of Speech and Language Therapy
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No